CLINICAL TRIAL: NCT00926926
Title: Effect of Oxybutynin Chloride Topical Gel on Gastric Emptying, Using the Acetaminophen Absorption Test
Brief Title: Effects of Oxybutynin Topical Gel on Gastric Emptying
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OTG0901
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
Keywords: Healthy volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active OTG (Experimental)
  Interventions: Drug: Oxybutynin Chloride Gel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Gel

INTERVENTIONS:
Drug: Oxybutynin Chloride Gel — Once daily for 7 days, followed by single dose of acetaminophen
  Arms: Active OTG
Drug: Placebo Gel — Once daily for 7 days, followed by single dose of acetaminophen
  Arms: Placebo

SUMMARY:
This study explores the effect of oxybutynin topical gel on gastric emptying

ELIGIBILITY:
Inclusion Criteria:

* Adult, healthy, post-menopausal females

Exclusion Criteria:

* Patients for whom OTG or acetaminophen is contraindicated.
* Abnormality of the GI tract.
* Taking drugs that affect gastric motility.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The effect of oxybutynin chloride topical gel administration on gastric emptying will be assessed by comparing the single dose relative bioavailability of acetaminophen | After 7 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Scott Olsen, MPH, Study Director — Watson Laboratories
Locations (1):
- Saint Charles, Missouri, United States